CLINICAL TRIAL: NCT00649298
Title: ACTIVE Dialysis - A Multicentre, Unblinded, Randomised, Controlled Trial to Assess Quality of Life, Clinical Outcomes and Cost Utility for Extended vs Standard Duration of Dialysis in Patients With End Stage Kidney Disease.
Brief Title: A Clinical Trial of IntensiVE Dialysis
Acronym: ACTIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GI-R-A001- 09
Record Dates: First submitted 2008-03-25; First posted 2008-04-01 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Renal Replacement Therapy; Renal Dialysis; End Stage Kidney Disease; End Stage Renal Disease; Uremia
Keywords: Randomized Controlled Trial; Clinical Trial; Controlled Clinical Trial; Clinical Trial, Phase IV; Multicenter Study; End Stage Kidney Disease; Hemodialysis; Renal Dialysis; Renal Replacement Therapy; Nocturnal Dialysis; Extended dialysis; Quality of Life; Quality Adjusted Life Year; Hypertrophy, Left Ventricular; Blood Pressure; Hypertension; Anemia; Hematinics; Erythropoiesis Stimulating Agents; Cost-utility Analysis; Economic Evaluation; Health Care Utilisation; Health Care Costs; Health Expenditures; Hospitalization; Cost Analysis; Cardiovascular Diseases; Acute Coronary Syndrome; Myocardial Infarction; Stroke; Cerebrovascular Disorders; Mortality; Arteriovenous Fistula; Arteriovenous Shunt, Surgical; Thrombosis; Infection
MeSH Terms: conditions — Kidney Failure, Chronic; Uremia; Hypertrophy, Left Ventricular; Hypertension; Anemia; Cardiovascular Diseases; Acute Coronary Syndrome; Myocardial Infarction; Stroke; Cerebrovascular Disorders; Arteriovenous Fistula; Thrombosis; Infections | interventions — Dialysis; Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extended hours (Experimental): 24 or more hours per week of hemodialysis
  Interventions: Procedure: haemodialysis
- standard hours (Active Comparator): 18 or less hours per week of hemodialysis
  Interventions: Procedure: haemodialysis

INTERVENTIONS:
Procedure: haemodialysis — Comparison of different weekly duration of haemodialysis treatment
  Other Names: Dialysis; Renal replacement therapy

SUMMARY:
This study will assess clinical outcomes of extended weekly hours of haemodialysis (>= 24 hours per week) compared with standard hours of haemodialysis (<=18 hours/week) in people with ESKD.

DETAILED DESCRIPTION:
A rapidly increasing volume of observational data suggests substantial benefits may be associated with an increased duration of dialysis. As well as improved quality of life, improved functioning and beneficial changes in a variety of laboratory parameters, it has been suggested that extended dialysis sessions might reduce mortality and major morbidity. Uncontrolled data from centres that have been providing extended dialysis shows dramatically lower mortality rates compared to those observed in centres providing standard duration dialysis. Recent analyses of extended dialysis conclude that the savings achieved in drug and hospitalization costs may lead to an overall reduction in costs compared with traditional forms of dialysis.

In this trial, we propose to examine the effects of extended dialysis (24 hours weekly or more) compared to standard dialysis (18 hours or less weekly) in patients with ESKD. The proposed study is a multi-centre, open label, randomised, controlled trial.

The study began with a pilot phase which was converted to the current main study on the receipt of peer-reviewed funding for the full study.

ELIGIBILITY:
Inclusion Criteria:

1. Incident or prevalent patients requiring maintenance haemodialysis therapy for ESKD
2. Aged 18 years or older
3. Undergoing dialysis for 18 hours per week or less
4. Suitable for either extended or standard dialysis in the view of the treating physician
5. Agreeable to randomisation

Exclusion Criteria:

1. Life expectancy of less than 6 months
2. Definite plans to undergo renal transplantation within 12 months of entry to the study
3. Inability to complete quality of life questionnaire
4. Concomitant major illness that would limit assessments and followup
5. High chance that the patient will not adhere to study treatment and follow up in the view of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary end-point for this study is the difference in the change in quality of life between the two groups from randomisation to the 12 month follow-up as measured by the EQ-5D instrument. | 12 months from randomisation

SECONDARY OUTCOMES:
Survival and cardiovascular analyses | 12 months
Quality of life and patient acceptability | 12 months
Safety outcomes | 12 months
Costs associated with each intervention | 12 months
Changes in biochemical and haematological parameters | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vlado Perkovic, MBBS PhD, Principal Investigator — The George Institute
Locations (40):
- Australia (14):
  - The Canberra Hospital, Canberra, Australian Capital Territory
  - RPAH/Concord, Sydney, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Sydney Dialysis Centre, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Gold Coast Hospital, Gold Coast, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Austin Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Canada (3):
  - UBC, Vancouver, British Columbia
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
- China (21):
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Civil Aviation General Hospital, Chaoyang District,, Beijing Municipality
  - China-Japan Friendship Hospital, Chaoyang District, Beijing Municipality
  - First Affiliated Hospital of Chinese PLA General Hospital, Haidian District, Beijing Municipality
  - Beijing Hospital, Xicheng District, Beijing Municipality
  - Peking University First Hospital, Xicheng District, Beijing Municipality
  - Peking University People's Hospital, Xicheng District, Beijing Municipality
  - Shenzhen Hospital of Peking University, Shenzhen, Guangdong
  - Fourth Hospital Affiliated to Hebei Medical University, Shijiazhuang, Hebei
  - Shijiazhuang First People's Hospital, Shijiazhuang, Hebei
  - Third Hospital Affiliated to Hebei Medical University, Shijiazhuang, Hebei
  - Zhengzhou University affiliated first hospital, Zhengzhou, Henan
  - First Affiliated Hospital of Inner Mongolia, Baotou Medical College, Baotou, Inner Mongolia
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Fourth Hospital Affiliated to Jilin University (FAW General Hospital), Changchun, Jilin
  - Dalian Medical affiliated first hospital, Dalian, Liaoning
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - The Chinese PLA Shanghai 85th Hospital, Shanghai, Shanghai Municipality
  - The second affiliated hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Huaxi Hospital of Sichuan University, Chengdu, Sichuan
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Auckland

REFERENCES:
- [Background] Jardine MJ, Zuo LI, Gray NA, de Zoysa J, Chan CT, Gallagher MP, Howard K, Hertier S, Cass A, Perkovic V; ACTIVE Dialysis Steering Committee. Design and participant baseline characteristics of 'A Clinical Trial of IntensiVE Dialysis': the ACTIVE Dialysis Study. Nephrology (Carlton). 2015 Apr;20(4):257-65. doi: 10.1111/nep.12385. PMID 25529309
- [Result] Smyth B, van den Broek-Best O, Hong D, Howard K, Rogers K, Zuo L, Gray NA, de Zoysa JR, Chan CT, Lin H, Zhang L, Xu J, Cass A, Gallagher M, Perkovic V, Jardine M. Varying Association of Extended Hours Dialysis with Quality of Life. Clin J Am Soc Nephrol. 2019 Dec 6;14(12):1751-1762. doi: 10.2215/CJN.06800619. Epub 2019 Oct 31. PMID 31672793
- [Result] Jardine MJ, Zuo L, Gray NA, de Zoysa JR, Chan CT, Gallagher MP, Monaghan H, Grieve SM, Puranik R, Lin H, Eris JM, Zhang L, Xu J, Howard K, Lo S, Cass A, Perkovic V; ACTIVE Dialysis Steering Committee; Paul. A Trial of Extending Hemodialysis Hours and Quality of Life. J Am Soc Nephrol. 2017 Jun;28(6):1898-1911. doi: 10.1681/ASN.2015111225. Epub 2017 Feb 1. PMID 28151412
- [Result] Zhan Z, Smyth B, Toussaint ND, Gray NA, Zuo L, de Zoysa JR, Chan CT, Jin C, Scaria A, Hawley CM, Perkovic V, Jardine MJ, Zhang L. Effect of extended hours dialysis on markers of chronic kidney disease-mineral and bone disorder in the ACTIVE Dialysis study. BMC Nephrol. 2019 Jul 12;20(1):258. doi: 10.1186/s12882-019-1438-3. PMID 31299919
- [Result] Liao JL, van den Broek-Best O, Smyth B, Hong D, Vo K, Zuo L, Gray NA, Chan CT, de Zoysa J, Perkovic V, Jiang L, Jardine M. Effect of extended hours dialysis on sleep quality in a randomized trial. Nephrology (Carlton). 2019 Apr;24(4):430-437. doi: 10.1111/nep.13236. PMID 29424935
- [Result] Gray NA, Zuo L, Hong D, Smyth B, Jun M, De Zoysa J, Vo K, Howard K, Wang J, Lu C, Liu Z, Cass A, Perkovic V, Jardine M. Quality of life in caregivers compared with dialysis recipients: The Co-ACTIVE sub-study of the ACTIVE dialysis trial. Nephrology (Carlton). 2019 Oct;24(10):1056-1063. doi: 10.1111/nep.13530. Epub 2019 Apr 29. PMID 30723975
- [Derived] Badve SV, Hawley CM, Johnson DW. Frequent versus standard hemodialysis. N Engl J Med. 2011 Mar 10;364(10):975; author reply 976. doi: 10.1056/NEJMc1100105. No abstract available. PMID 21388319